CLINICAL TRIAL: NCT00000375
Title: Continuation ECT Vs Pharmacotherapy--Efficacy And Safety
Brief Title: Continuation Electroconvulsive Therapy Vs Medication to Prevent Relapses in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: MH55495; NCT00069394 (obsolete NCT alias)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2005-12

CONDITIONS: Major Depressive Disorder
Keywords: Adult; Antidepressive Agents; Depressive Disorder; Electroconvulsive Therapy; Female; Human; Lithium; Male; Nortriptyline; Serotonin Uptake Inhibitors; Antidepressive Agents -- *therapeutic use; Antidepressive Agents -- adverse effects; Lithium -- *therapeutic use; Lithium -- adverse effects; Nortriptyline -- *therapeutic use; Nortriptyline -- adverse effects
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder

INTERVENTIONS:
Drug: Nortriptyline-lithium (NOR-Li)
Procedure: Bilateral electroconvulsive therapy (ECT)
Drug: Continuation therapy
Behavioral: Continuation ECT

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of two treatments to prevent relapses in seriously ill patients with major depressive disorder (MDD) who have responded to electroconvulsive therapy (ECT). Patients will either continue to receive ECT (continuation electroconvulsive therapy [C-ECT]), or they will be treated with antidepressant medications.

ECT is a highly effective treatment for MDD; however, relapses are a major concern. To prevent relapse in patients who have responded to ECT, the common treatment is antidepressants as continuation therapy (following the initial therapy in order to continue treating the disorder). Relapses, however, can still occur even after antidepressant continuation therapy. This study will evaluate a potent antidepressant combination in order to prevent relapse. C-ECT is another option that needs to be tested.

If the patient responds to the first round of ECT, he/she will be assigned randomly (like tossing a coin) to either continue receiving ECT or to receive an antidepressant combination of nortriptyline plus lithium (NOR-Li) for 6 months. The patient will have psychological tests before, shortly after, and 3 months after the first round of ECT, and at the end of the 6-month continuation trial. Patients will be monitored for symptoms and side effects. All patients will have urine tests to test for drug abuse.

An individual may be eligible for this study if he/she:

Has major depressive disorder and responds positively to ECT treatment and is 18 to 80 years old.

DETAILED DESCRIPTION:
To define the role of continuation electroconvulsive therapy (C-ECT) in relapse-prevention of seriously ill patients with major depressive disorder (MDD). To determine the relative efficacy and safety of C-ECT in comparison to the traditional approach of continuation pharmacotherapy (C-PHARM) to prevent relapses of MDD.

Electroconvulsive therapy (ECT) is a highly effective treatment for MDD that is helpful for patients with the most severe forms of affective illness; however, relapse after successful acute phase ECT or pharmacotherapy remains a major public health problem. To prevent relapse in patients with MDD who have responded to ECT, the common practice is to prescribe an antidepressant (e.g., a tricyclic [TCA], a selective serotonin reuptake inhibitor [SSRI], or lithium) as continuation therapy. Recent studies show an alarmingly high relapse rate after ECT despite conventional continuation pharmacotherapy (C-PHARM). Continuation ECT (C-ECT) is also in widespread clinical use; however, its efficacy and safety have never been rigorously tested.

Investigators at four sites (Mayo Clinic, UMDNJ-New Jersey Medical School, Zucker Hillside Hospital, and University of Texas SW Medical Center, Dallas) randomize patients to receive either C-ECT or an aggressive pharmacological strategy (nortriptyline and lithium in combination, [NOR-Li]) for 6 months following response to acute phase ECT. Raters at each site evaluate symptoms and side effects. On the basis of edited videotapes obtained at regular intervals, a site-independent, blinded evaluator also assesses symptoms. A neuropsychological battery is administered prior to acute phase ECT, shortly after the ECT course, 3 months after the end of the acute phase treatment, and at the end of the 6-month continuation trial. These continuation therapies are compared in their effects on relapse, cognitive performance, global functioning, side effects, and perceived health status. NOR and Li levels are optimized by blood level monitoring. Bilateral ECT, at progressively increasing intervals, are used for C-ECT. Methods are included to ensure the integrity of clinical diagnoses, symptom severity assessment, data collection and entry, and treatment delivery. In all patients, surreptitious use of prescription or recreational drugs is monitored by urine testing.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Major depressive disorder that is responsive to acute phase ECT.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-02

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kellner, MD, Study Chair; Mustafa Husain, MD, Principal Investigator; Teresa Rummans, MD, Principal Investigator; George Petrides, Principal Investigator
Locations (1):
- New Jersey Medical School, Newark, New Jersey, United States

REFERENCES:
- [Derived] Husain MM, McClintock SM, Rush AJ, Knapp RG, Fink M, Rummans TA, Rasmussen K, Claassen C, Petrides G, Biggs MM, Mueller M, Sampson S, Bailine SH, Lisanby SH, Kellner CH. The efficacy of acute electroconvulsive therapy in atypical depression. J Clin Psychiatry. 2008 Mar;69(3):406-11. doi: 10.4088/jcp.v69n0310. PMID 18278988